CLINICAL TRIAL: NCT04864418
Title: A Phase 1 Study to Evaluate the Safety, Tolerability and Optimal Immunogenic Dose of Therapeutic Cancer Vaccine (AST-021p) in Patients With Advanced Solid Tumors
Brief Title: AST-021p Study in Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aston Sci. Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PN-021-11
Record Dates: First submitted 2021-04-22; First posted 2021-04-28 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-02

CONDITIONS: Advanced Cancer
Keywords: cancer vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Cohort group of AST-021p for dose-escalation (Experimental): 4 cohort groups for AST- 021p administration:
  Group 1) 1.2mg AST-021p, Montanide ISA 51 VG and rhuGM-CSF
  Group 2) 2.4mg AST-021p, Montanide ISA 51 VG and rhuGM-CSF
  Group 3) 3.6mg AST-021p, Montanide ISA 51 VG and rhuGM-CSF
  Group 4) 4.8mg AST- 021p, Montanide ISA 51 VG and rhuGM-CSF
  Interventions: Drug: AST-021p

INTERVENTIONS:
Drug: AST-021p — 3 priming immunization (2weeks x3) in 4 cohort groups (1.2mg, 2.4mg, 3.6mg and 4.8mg AST-021p) if possible, 3 boosting immunization (4weeks x 3) in cohort groups after priming immunization

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability and optimal Immunogenic dose of therapeutic cancer vaccine (AST-021p) in patients With advanced solid tumors

A phase 1 study

DETAILED DESCRIPTION:
Recurrent or advanced solid cancer patients without applicable standard treatments will be included in the 4 dose groups (4 cohort groups- 1.2mg, 2.4mg,3.6mg and 4.8mg) of AST-021p. Participants in each cohort group will be treated 3 times in each dose (3 priming immunications)

This study will apply a modified 3+3 design for dose-escalation.

1 participant will be registered in the lowest dose cohort group(1.2mg) and when the safety and tolerance of the AST-021p(1.2mg) are identified in the the first group, dose will be increased sequentially and accordingly, the safety and tolerance will be assessed for six participants in the other cohort groups (group2(2.4mg), group3(3.6mg) and group4(4.8mg)).

Participants receiving priming immunization only will be assessed up to End of Treatment(EOT) and participants who recive boosting immunization will be evaluated until the end of study(EOS).

ELIGIBILITY:
Inclusion Criteria:

* has recurrent or metastatic solid cancer that has been proven histologically or cytologically and cannot be treated with surgery or radiotherapy for the purpos of complete remission
* does not have a standard treatment that can be applied clinically according to the investigator's judgment
* has an expected life expectancy of more than 3 months
* adults aged 19 or older based on screening day
* ECOG performance status : 0~1

Exclusion Criteria:

* Has a history of hypersensitivity or other contraindications to rhGM-CSF and Montanide ISA 51 VG
* Has a history of other primary malignant tumor
* Has autoimmune diseases or inflammatory diseases
* Has a history of active primary immunodeficiency disease
* Has active infection including tuberculosis, hepatitis B, hepatitis C or human immunodeficiency virus (HIV) infection
* Is pregnant or breastfeeding or expecting to conceive children
* has a history of immune suppression therapy ≤4 weeks prior to the screening day

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by AST-021p | 6weeks after AST-021p administration in each cohort group
  After AST-021p administration in patients with advance solid tumor, safety and tolerance are assessed for each dose group(1.2mg,2.4mg, 3.6mg &4.8mg)
  Safety and tolerance evaluation variables :
  1)adverse events 2) Vital signs 3)Physical examination 4) ECOG performance evaluation 5)ECG examination 6)Laboratory examination

SECONDARY OUTCOMES:
Immunogenicity assessment | 8weeks after ASP-021p administration (Priming immunization case) or 20weeks after ASP-021p(Priming immunization and Boosting immunization case)
  ASP-021p specific IFN-γ ELISpot(Interferon Gamma Enzyme-linked immunospot) test results and ASP-021p4 & ASP-021p5 specific IFN-γ ELISpot ( spots/250,000 Tcell of pre ASP-021p and post ASP-021p)
Tumor response assessment | Overall study period approximately up to 5months
  Disease control rate (%), objective response rate(%) and duration of response (days & weeks)
Progression-Free Survival rate | Overall study period approximately up to 5months
  PFS rate (%) at End of Study
Overall Survival rate | Overall study period approximately up to 5months
  OS rate (%) at End of study

CONTACTS AND LOCATIONS:
Overall Officials: Kyong Hwa Park, MD. PhD, Principal Investigator — Korea University Anam Hospital
Locations (3):
- South Korea (3):
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul ST. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No